CLINICAL TRIAL: NCT02617953
Title: Variable Changes in Continuous Resting EEG(Electroencephalography) and Auditory ERP(Event-related Potential) Before and After Transcranial Magnetic Stimulation Treatment; Double Blind Randomized Controll Trails
Brief Title: Objective Diagnosis Method and Efficacy of Repetitive Transcranial Magnetic Stimulation as a Treatment for Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-199-08-14
Record Dates: First submitted 2015-10-28; First posted 2015-12-01 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Tinnitus
Keywords: Tinnitus; EEG; ERP
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active rTMS(A) (Experimental): low frequency frontal and temporal repetitive transcranial magnetic stimulation
  Interventions: Device: Active rTMS(A)
- Active rTMS(B) (Experimental): Temporal low frequency repetitive transcranial magnetic stimulation
  Interventions: Device: Active rTMS(B)
- Sham condition(C) (Sham Comparator): low frequency frontal and temporal repetitive transcranial magnetic stimulation
  Interventions: Device: Sham condition(C)

INTERVENTIONS:
Device: Active rTMS(A) — repetitive transcranial magnetic stimulation:1000 stimuli of 1Hz rTMS over the left dorsolateral prefrontal cortex followed by 2000 stimuli of 1 Hz rTMS over the left primary auditory cortex , each consisting of 4 days of rTMS treatment.
  auditory ERP,continuous resting EEG and MRI are measured pre-treatment rTMS and auditory ERP,continuous resting EEG are measured two weeks after rTMS treatment. Tinnitus subjects were asked to perform an interval duration paried pulse task before and after the rTMS train.
  Arms: Active rTMS(A)
Device: Active rTMS(B) — repetitive transcranial magnetic stimulation:1000 stimuli of 1Hz rTMS over the left dorsolateral prefrontal cortex followed by 2000 stimuli of 1 Hz rTMS over the left primary auditory cortex , each consisting of 4 days of rTMS treatment.
  auditory ERP,continuous resting EEG and MRI are measured pre-treatment rTMS and auditory ERP,continuous resting EEG are measured two weeks after rTMS treatment. Tinnitus subjects were asked to perform an interval duration paried pulse task before and after the rTMS train.
  Arms: Active rTMS(B)
Device: Sham condition(C) — The sham stimulation looks and sounds like the active coil, but diverts the magnetic field away from the patient.
  auditory ERP,continuous resting EEG and MRI are measured pre-treatment rTMS and auditory ERP,continuous resting EEG are measured two weeks after rTMS treatment. Tinnitus subjects were asked to perform an interval duration paried pulse task before and after the rTMS train.
  Arms: Sham condition(C)

SUMMARY:
Investigation of objective tinnitus diagnosis method through measurement of continuous resting EEG, auditory ERP before and after Repetitive Transcranial Magnetic Stimulation (rTMS) treatment of tinnitus.

DETAILED DESCRIPTION:
Tinnitus is defined as the subjective perception of a sound in the absence of any physical sound. Therefore, accurate diagnosis of tinnitus is so difficult.

So, Investigators measure auditory ERP through autonomously developed system to make a objective diagnosis tinnitus. Moreover, patients undergo continuous resting EEG measurement.

In this study investigators examined the efficacy of rTMS treatment for tinnitus and check into changes in brain connectivity or auditory task with ERP, continuous resting EEG before and after rTMS. And develop a new test that can detect tinnitus objectively in humans, using the prepulse gap paradigm

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic tinnitus
* Chronic subjective tinnitus for more than 6 months
* Subject is naive regarding rTMS
* Other concurrent treatments: A four-week washout from any other tinnitus treatment or management program is required prior to entering this study
* Stable enough to complete this study per the opinion of the Study Physician
* No restrictions, provided the dosages have been in place for at least 3 months
* A three month washout from any other tinnitus treatment or management program is required prior to entering this study.

Exclusion Criteria:

* Objective tinnitus or tinnitus with treatable cause
* Presence of intracranial or intraocular ferromagnetic materiel or particles
* Cardiac pacemaker or other electronic implants (including cochlear implant) Serious heart disease or other unstable major medical condition
* Personal history of central nervous system disorder, head injury, stroke or seizures
* Familial history of epilepsy
* Concomitant medication with antidepressants and antipsychotics
* Pregnant women
* Others known contraindications to rTMS or brain MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change of Tinnitus Handicap Inventory (THI) before and after treatment , difference in brain gating and connectivity before and after treatment. | Change from Baseline THI at 6 months

SECONDARY OUTCOMES:
Change of Visual Analogue Scale (VAS) for tinnitus states before and after treatment. | Change from Baseline VAS at 6 months
Positive And Negative Affect Schedule(PANAS) | Baseline, 1, 2 and 3 month after the first intervention
Beck's Depression Inventory (BDI) | Baseline
State-Trait Anxiety Inventory (STAI) | Baseline
Pittsburgh Sleep Quality Index (PSQI) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Whan Suh, MD, ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No